CLINICAL TRIAL: NCT05156047
Title: A Double-Blind, Placebo-Controlled, Randomized Withdrawal Study to Evaluate the Safety and Efficacy of Pitolisant in Adult Patients With Idiopathic Hypersomnia
Brief Title: A Phase 3 Study to Assess the Safety and Efficacy of Pitolisant in Adult Patients With Idiopathic Hypersomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HBS-101-CL-010
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Idiopathic Hypersomnia
Keywords: pitolisant; histamine; sleepiness
MeSH Terms: conditions — Idiopathic Hypersomnia; Sleepiness

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized withdrawal
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-blind pitolisant (Active Comparator): Double-blind pitolisant administered once daily in the morning upon wakening for 4 weeks during the Double-Blind Randomized Withdrawal Phase
  Interventions: Drug: Double-blind pitolisant
- Double-blind placebo (Placebo Comparator): Matching placebo administered once daily in the morning upon wakening for 4 weeks during the Double-Blind Randomized Withdrawal Phase
  Interventions: Drug: Double-blind placebo
- Open-label pitolisant (Experimental): Open-label pitolisant administered once daily in the morning upon wakening for 8 weeks during the Open-Label Phase
  Interventions: Drug: Open-label pitolisant

INTERVENTIONS:
Drug: Open-label pitolisant — Pitolisant 4.45 mg tablets: white, round, plain, biconvex film-coated tablet, 3.7 mm in diameter. Each tablet contains 5 mg of pitolisant hydrochloride equivalent to 4.45 mg of pitolisant.
  Pitolisant 17.8 mg tablets: white, round, plain, biconvex film-coated tablet, 7.5 mm in diameter. Each tablet contains 20 mg of pitolisant hydrochloride equivalent to 17.8 mg of pitolisant.
  Arms: Open-label pitolisant
Drug: Double-blind placebo — Matching placebo tablets will be provided for each strength of active pitolisant film-coated tablets.
  Arms: Double-blind placebo
Drug: Double-blind pitolisant — Pitolisant 4.45 mg tablets: white, round, plain, biconvex film-coated tablet, 3.7 mm in diameter. Each tablet contains 5 mg of pitolisant hydrochloride equivalent to 4.45 mg of pitolisant.
  Pitolisant 17.8 mg tablets: white, round, plain, biconvex film-coated tablet, 7.5 mm in diameter. Each tablet contains 20 mg of pitolisant hydrochloride equivalent to 17.8 mg of pitolisant.
  Arms: Double-blind pitolisant

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of pitolisant compared with placebo in treating excessive daytime sleepiness (EDS) in patients with idiopathic hypersomnia (IH) age ≥18 years.

Key secondary objectives of this study are to assess the impact of pitolisant on:

* Overall symptoms of IH
* Patient impression of overall change in their symptoms of IH
* Investigator assessment of overall disease severity of IH

Other secondary objectives of this study are to assess the impact of pitolisant in patients with IH on:

* Patient impression of overall severity of their EDS
* Functional status and activities of daily living
* Sleep-related impairment
* Sleep inertia
* Cognitive function

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized withdrawal study in adult patients (ages ≥18 years) with IH. The study will consist of a Screening Period (up to 28 days), an 8-week Open-Label Phase, and a 4-week Double-Blind Randomized Withdrawal Phase.

The Open-Label Phase of the study will be 8 weeks, which includes a 6-week Dose Optimization Period and a 2-week Stable Dose Period. In the Dose Optimization Period, all patients will be titrated to their optimal dose of open-label pitolisant (17.8 mg or 35.6 mg) based on Investigator assessment of tolerability and efficacy. The 3-week titration period will be followed by 3 weeks of flexible dosing (weeks 4-6) during which patients will continue to receive their optimal dose of 17.8 mg or 35.6 mg open-label pitolisant. Patients taking a strong CYP2D6 inhibitor will be allowed in the study; however, for these patients, the maximum permitted daily dose of pitolisant will be 17.8 mg. Following completion of the 6-week Dose Optimization Period, patients will enter the 2-week Stable Dose Period. During this period, patients will remain at their optimal dose (the same dose they were taking at the end of the Dose Optimization Period [17.8 mg or 35.6 mg]) of open-label pitolisant for 2 weeks; dose adjustments are not allowed during the Stable Dose Period. At the end of the Stable Dose Period, patients will be defined as responders or non-responders. Responders will be randomized in a 1:1 ratio to receive blinded study drug (pitolisant or matching placebo) in the Double-Blind Randomized Withdrawal Phase of the study. Non-responders will not be randomized to treatment in the Double-Blind Randomized Withdrawal Phase and will complete two safety follow-up telephone contacts (TCs) at 15 (±3) days and 30 (+3) days after their final dose of open-label pitolisant.

During the Double-Blind Randomized Withdrawal Phase, patients (approximately 64 patients per treatment group) will receive blinded study drug either at the same dose they were taking in the Stable Dose Period (17.8 mg or 35.6 mg pitolisant) or matching placebo. The duration of the Double-Blind Randomized Withdrawal Phase will be 4 weeks (weeks 9-12); dose adjustments are not permitted during this phase of the study. After completion of the Double-Blind Randomized Withdrawal Phase (End-of Treatment [EOT] Visit is on Day 84, the last day of blinded treatment), patients will complete two safety follow-up TCs with the site at 15 (±3) days and 30 (+3) days after their final dose of blinded study drug, which will include assessment for AEs and concomitant medication use; alternatively, patients will have the opportunity to enroll in a long-term, open-label safety study under a separate protocol. Patients who opt to enroll into the long-term, open-label study will not complete the 15 day and 30 day follow-up TCs.

ELIGIBILITY:
Inclusion Criteria:

1. Is able to provide voluntary, written informed consent.
2. Has a current diagnosis of IH per International Classification of Sleep Disorders Third Edition (ICSD 3) criteria.
3. Male or female patient age ≥18 years at the time of Screening.
4. Has an ESS score of ≥12 at Screening and at Baseline (Visit 2).
5. Has a PGI-S score of moderate, severe, or very severe at Screening and at Baseline (Visit 2).
6. For patients being treated for OSA or other hypoventilatory conditions, patients must be compliant as demonstrated by BiPAP/CPAP therapy with 30 days of data showing ≥4 hours of BiPAP/CPAP therapy per night for ≥70% of nights. If not on BiPAP/CPAP therapy, patients being treated for OSA must be compliant as determined by the Investigator with their medical device or oral appliance. Data must be from within 90 days prior to the Screening visit. Patients must agree to maintain compliance with their treatment for OSA throughout the duration of the study.
7. If on a treatment that could affect daytime sleepiness (including but not limited to oxybates, stimulants, modafinil, and armodafinil):

   1. Must be on a stable dose for at least 2 months prior to Screening and agree to continue the stable dose for the duration of the study.
   2. If not on a stable dose for 2 months prior to Screening, washout for 5 half-lives or 14 days, whichever is longer, prior to Day 1 and agree to remain off these treatments until completion of the study.
8. A patient who is a female of child-bearing potential (FCBP) must have a negative serum pregnancy test at the Screening Visit and negative urine pregnancy test at the Baseline Visit (Visit 2) and at the end of the Stable Dose Period (Visit 4) and agree to remain abstinent or use an effective method of non-hormonal contraception to prevent pregnancy for the duration of the study and for 21 days after final dose of study drug.
9. Must have a negative result on urine drug screen at the Screening Visit, Baseline Visit (Visit 2) and at the end of the Stable Dose Period (Visit 4), except for medications that are prescribed by a healthcare provider for medical conditions.
10. In the opinion of the Investigator, the patient is capable of understanding and complying with the protocol and administration of oral study drug.

Exclusion Criteria:

1. Has hypersomnia due to another medical disorder (e.g., narcolepsy).
2. Has an AHI of ≥10 as determined by the most recent sleep study or BiPAP/CPAP device readout.
3. Has a clinically significant hypoventilatory condition as determined by the Investigator.
4. Has a primary diagnosis of a psychiatric illness that is not well controlled.
5. Patients taking antidepressants who have not been on a stable dose of their antidepressant for at least 12 weeks prior to Screening; patients on a stable dose of their antidepressant for at least 12 weeks prior to Screening must agree to continue their stable dose for the duration of the study.
6. Experiences a mean of <6 hours of sleep per night based on sleep diary during Screening (patients need to record at least 7 nights within a 10-day period in their sleep diary within 14-days prior to the Baseline Visit [Visit 2]).
7. Consistently consumes >600 mg of caffeine per day and is unable/unwilling to reduce caffeine intake to ≤600 mg per day for the duration of the study.
8. Does not agree to discontinue any prohibited medication or substance listed in the protocol.
9. Is currently or has previously used pitolisant.
10. Is currently breastfeeding or planning to breastfeed over the course of the study. Lactating women must agree not to breastfeed for the duration of the study and for 21 days after final dose of study drug.
11. Participation in an interventional research study involving another investigational medication, device, or behavioral treatment within 28 days or within 5 half-lives of the investigational medication (whichever is longer) prior to Screening.
12. Has a diagnosis of ESRD (estimated glomerular filtration rate [eGFR] of <15 mL/minute/1.73 m²) or severe hepatic impairment (Child-Pugh C).
13. Has a diagnosis of moderate or severe renal impairment (eGFR ≥15 to ≤59 mL/minute/1.73 m²) or moderate hepatic impairment (Child-Pugh B) at Screening or at any time during the study.
14. Has a history of long corrected QT interval (QTc) syndrome or corrected QT interval using Fridericia's formula (QTcF) >450 msec for males or >470 msec for females (QTcF = QT / 3√ RR) at Screening.
15. Is receiving and is unable to discontinue a medication known to prolong the QT interval.
16. Is receiving a concomitant medication that is known to be a strong CYP3A4 inducer, or a centrally acting histamine 1 (H1) receptor antagonist; patients who undergo a washout of these medications of at least 5 half-lives or one week (whichever is longer) may be enrolled in the study. Use of strong CYP2D6 inhibitors is allowed; however, for these patients the maximum permitted daily dose of pitolisant is 17.8 mg.
17. Is a known CYP2D6 poor metabolizer (PM).
18. Has abnormal laboratory values at Screening that are clinically significant as determined by the Investigator.
19. Has initiated any new or change in allied health therapies or interventions that can interfere with the study outcomes within 28 days prior to Screening and at any time during the study, based on the Investigator's judgment.
20. Has a current or recent (within 1 year) history of a substance use disorder or dependence disorder, including alcohol, tobacco, and caffeine use disorders as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).
21. Has planned surgery during the study.
22. Has a significant risk of committing suicide or suicidality based on history; routine psychiatric examination; Investigator's judgment; or an answer of "yes" on any question other than questions 1 to 3 (for the previous month) or "yes" on any question in the suicidal behavior section (for the past year) of the Columbia-Suicide Severity Scale (C-SSRS), Baseline/Screening.
23. Based on the judgment of the Investigator, is unsuitable for the study for any reason, including but not limited to an unstable or uncontrolled medical condition or one that might interfere with the conduct of the study, confound interpretation of study results, pose a health risk to the patient, or compromise the integrity of the study. This exclusion criterion applies not only to entry into the study, but also to continuation in the study, should such an unstable, uncontrolled, or serious medical condition arise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Excessive Daytime Sleepiness | Week 8 to Week 12
  Change in Epworth Sleepiness Scale score from the end of the Stable Dose Period to the end of the 4-week Double-Blind Randomized Withdrawal Phase for pitolisant compared with placebo.
  The score of the Epworth Sleepiness Scale ranges from 0 to 24. A decrease in score represents an improvement in excessive daytime sleepiness.

SECONDARY OUTCOMES:
Symptoms of idiopathic hypersomnia | Week 8 to Week 12
  Change in Idiopathic Hypersomnia Severity Scale.
  The score of the Idiopathic Hypersomnia Severity Scale ranges from 0 to 50. A decrease in score represents an improvement in symptoms of idiopathic hypersomnia.
Symptoms of idiopathic hypersomnia | Week 8 to Week 12
  Percent of patients who worsen on the Patient Global Impression of Change.
  The Patient Global Impression of Change is a five item scale that ranges from much better to much worse. An assessment of being better represents an improvement in the patient's overall perception of the change in their idiopathic hypersomnia.
Symptoms of idiopathic hypersomnia | Week 8 to Week 12
  Change in Clinical Global Impression of Severity.
  The Clinical Global Impression of Severity is a five item scale that ranges from none to very severe. An assessment of less severe symptoms represents an improvement in the clinician's perception of the patient's overall clinical status related to idiopathic hypersomnia.
Symptoms of idiopathic hypersomnia | Week 8 to Week 12
  Change in Patient Global Impression of Severity of their excessive daytime sleepiness.
  The Patient Global Impression of Severity is a five item scale that ranges from none to very severe. An assessment of less severe symptoms represents an improvement in the patient's perception of the severity of their excessive daytime sleepiness.
Functional outcomes of sleep | Week 8 to Week 12
  Change in Functional Outcomes of Sleep Questionnaire 10-item Version.
  The score of the Functional Outcomes of Sleep Questionnaire 10-item Version ranges from 5 to 20. An increase in score represents an improvement in the patient's impression of the impact of hypersomnia on multiple activities of everyday living.
Sleep related impairments during wakefulness | Week 8 to Week 12
  Change in Patient-Reported Outcomes Measurement Information System, Sleep-Related Impairment.
  The score of the Patient-Reported Outcomes Measurement Information System, Sleep-Related Impairment ranges from 8 to 40. A decrease in score represents an improvement in the patient's impression of the impact of hypersomnia on multiple activities of everyday living.
Sleep inertia | Week 8 to Week 12
  Change in Sleep Inertia Questionnaire.
  The Sleep Inertia Questionnaire ranges from 21 to 105. A decrease in score represents an improvement in the patient's ability to wake up after sleep.
Working Memory | Week 8 to Week 12
  Change in Cogstate One Back Test.
  The Cogstate One Back Test is a computerized test. A faster speed represents a better working memory test performance.
Attention | Week 8 to Week 12
  Change in Cogstate Identification Test.
  The Cogstate Identification Test is a computerized test. A faster speed represents an improvement in attention test performance.
Psychomotor Function | Week 8 to Week 12
  Change in Cogstate Detection Test.
  The Cogstate Detection Test is a computerized test. A faster speed represents an improvement in psychomotor test performance.

CONTACTS AND LOCATIONS:
Locations (58):
- United States (58):
  - Phoenix Medical Group, Peoria, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Cedars-Sinai Medical Towers, Los Angeles, California
  - University of California- Los Angeles, Los Angeles, California
  - Sleep Medicine Specialists of California, San Ramon, California
  - SDS Clinical Trials Inc., Santa Ana, California
  - Santa Monica Clinical Trials, Santa Monica, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Norwalk Hospital Sleep Center, Norwalk, Connecticut
  - Meris Clinical Research, Brandon, Florida
  - St. Francis Medical Institute, Clearwater, Florida
  - Sleep Medicine Specialists of South Florida, PA, Miami, Florida
  - Pasadena Center For Medical Research, LLC, St. Petersburg, Florida
  - Florida Pediatric Research Institute, Winter Park, Florida
  - Neurotrials Research Inc., Atlanta, Georgia
  - The Neurological Center of North GA, Gainesville, Georgia
  - Northwestern University, Chicago, Illinois
  - NorthShore Uni HealthSys-Glenbrook Hospital, Glenview, Illinois
  - OSF HealthCare Saint Francis Medical Center, Peoria, Illinois
  - Helene A. Emsellem MD PC, Chevy Chase, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Neurocare, INC, Newton, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - Bronson Sleep Health, Portage, Michigan
  - Clinical Neurophysiology Services, Sterling Heights, Michigan
  - Minnesota Lung Center, Edina, Minnesota
  - Minnesota Lung Center, Woodbury, Minnesota
  - St. Luke's Sleep Medicine and Research Center, Chesterfield, Missouri
  - Clayton Sleep Institute, St Louis, Missouri
  - Great Plains Health, North Platte, Nebraska
  - Neurology Specialists of Monmouth County, PA, West Long Branch, New Jersey
  - Northwell Health, New Hyde Park, New York
  - Research Carolina Elite LLC, Denver, North Carolina
  - Duke University School of Medicine, Durham, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - ARSM Research, Huntersville, North Carolina
  - NeuroScience Research Center, LLC, Canton, Ohio
  - Intrepid Research, LLC, Cincinnati, Ohio
  - Rainbow Babies Children's Hospital, Cleveland, Ohio
  - Cleveland Clinc, Cleveland, Ohio
  - Ohio Sleep Medicine and Neuroscience Institue, Dublin, Ohio
  - North Star Medical Research, Middleburg, Ohio
  - CardioVoyage, Ardmore, Oklahoma
  - Brian Abaluck, LLC, Paoli, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Respiratory Specialists, Wyomissing, Pennsylvania
  - Medical University of South Carolina- Institute of Psychiatry, Charleston, South Carolina
  - Bogan Sleep Consultants, Columbia, South Carolina
  - Lowcountry Lung Critical Care, North Charleston, South Carolina
  - Advanced Center for Sleep Disorders, Chattanooga, Tennessee
  - Neurology Clinic, P.C., Cordova, Tennessee
  - FutureSearch Trials of Neurology LP, Austin, Texas
  - Central Texas Neurology Consultants, PA, Round Rock, Texas
  - Comprehensive Sleep Medicine Associates, Sugar Land, Texas
  - Northwest Houston Neurology and Sleep, Tomball, Texas
  - Children's Hospital of the King's Daughter, Norfolk, Virginia
  - West Virginia University - Department of Neurology, Morgantown, West Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin